CLINICAL TRIAL: NCT01918059
Title: Prospective, Randomized, Controlled Trial of Tissue Adhesive (Octyl-2-Cyanoacrylate) vs. Traditional Suture in Traumatic Lid Laceration Repair
Brief Title: Cosmetic Outcome Study of Lid Laceration Repair With Suture Versus Tissue Adhesive
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment difficulties
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Judianne Kellaway, Clinical Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-13-0276
Record Dates: First submitted 2013-07-30; First posted 2013-08-07 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Eyelid Laceration
Keywords: Trauma; Eyelid; Laceration; Tissue adhesive; suture; cosmetic; octyl-2-cyanoacrylate
MeSH Terms: conditions — Wounds and Injuries; Lacerations | interventions — octyl 2-cyanoacrylate; Cyanoacrylates; Tissue Adhesives; Polypropylenes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Non-absorbable suture skin closure (Experimental): The superficial eyelid skin will be repaired with simple interrupted sutures with non-absorbable suture (6-0 polypropylene) after repair of any deep component of the laceration.
  Interventions: Procedure: Non-absorbable suture skin closure
- Absorbable suture skin closure (Experimental): The superficial eyelid skin will be repaired with simple interrupted sutures with absorbable suture (surgical gut) after repair of any deep component of the laceration.
  Interventions: Procedure: Absorbable suture skin closure
- Tissue Adhesive skin closure (Experimental): The superficial eyelid skin will be repaired with layers of tissue adhesive (octyl-2-cyanoacrylate) after repair of any deep component of the laceration.
  Interventions: Procedure: Tissue Adhesive skin closure

INTERVENTIONS:
Procedure: Tissue Adhesive skin closure — The approach to repair will follow standard technique. If eyelid marginal component is present, margin repair will be performed with two 6-0 interrupted silk sutures: one at the gray line and one at the lash line. If the tarsus requires reapproximation, this will carefully be done using interrupted polyglactin vicryl sutures. The superficial skin will then be repaired with tissue adhesive (octyl-2-cyanoacrylate).
  Other Names: octyl-2-cyanoacrylate; cyanoacrylate; tissue adhesive
  Arms: Tissue Adhesive skin closure
Procedure: Absorbable suture skin closure — The approach to repair will follow standard technique. If eyelid marginal component is present, margin repair will be performed with two 6-0 interrupted silk sutures: one at the gray line and one at the lash line. If the tarsus requires reapproximation, this will carefully be done using interrupted polyglactin vicryl sutures. The superficial skin will then be repaired with absorbable sutures (surgical gut).
  Other Names: gut; surgical gut
  Arms: Absorbable suture skin closure
Procedure: Non-absorbable suture skin closure — The approach to repair will follow standard technique. If eyelid marginal component is present, margin repair will be performed with two 6-0 interrupted silk sutures: one at the gray line and one at the lash line. If the tarsus requires reapproximation, this will carefully be done using interrupted polyglactin vicryl sutures. The superficial skin will then be repaired with either non-absorbable sutures (6-0 polypropylene).
  Other Names: prolene; polypropylene
  Arms: Non-absorbable suture skin closure

SUMMARY:
This project is a randomized, controlled trial investigating wound cosmetic appearance after repair of traumatic lid lacerations with three different approaches to skin closure: absorbable sutures, non-absorbable sutures, and tissue adhesive. Photographs will be taken at two intervals after repair and later blindly assessed using standard cosmetic assessment scales. The investigators hypothesize that cosmetic wound outcome will be equivalent in across all three treatment arms.

DETAILED DESCRIPTION:
This project is a randomized, controlled trial investigating the cosmetic appearance after repair of traumatic lid lacerations with three different approaches to skin closure: absorbable sutures (surgical gut suture), non-absorbable sutures (polypropylene suture), and tissue adhesive (octyl-2-cyanoacrylate). The population will include patients presenting to Memorial Hermann Hospital requiring repair of traumatic lid lacerations. The study will include partial thickness, full-thickness, and margin-involving lacerations where first standard layered tarsal and marginal suture repair will be performed if necessary, and then the patient will be randomized to superficial skin closure with either polypropylene suture closure, surgical gut suture closure, or tissue adhesive closure. Subjects will be followed in an outpatient setting at 1 week and 1 month post-repair at which time standardized photographs will be taken and later assessed using two standardized appearance assessment tools: Visual Analogue Scale (VAS) and Hollander Wound Evaluation Score (HWES).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Any laceration caused by trauma and involving the skin of the upper and/or lower eyelid.
* Must be able to understand and sign an informed consent when applicable and Health Insurance Portability and Accountability Act(HIPAA) form that has been approved by an Institutional Review Board (IRB) or follow standard informed consent procedure of the IRB

Exclusion Criteria:

* Eyelid lacerations that include avulsion or missing eyelid tissue
* Patients with known hypersensitivity to octyl-2-cyanoacrylate or previous poor reaction to octyl-2-cyanoacrylate
* Eyelid lacerations resulting in necrosis or ischemia of tissue prior to repair
* Patients who demonstrate intoxication or mental status changes that would make them unfit to provide informed consent for repair

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Cosmetic wound appearance | 1 month after repair
  Cosmetic appearance will be assessed using two wound assessment methods: the Visual Analogue Scale (VAS) and the Hollander Wound Evaluation Scale (HWES).

CONTACTS AND LOCATIONS:
Overall Officials: Judianne Kellaway, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Memorial Hermann Hospital - Texas Medical Center, Houston, Texas, United States

REFERENCES:
- [Background] Singer AJ, Arora B, Dagum A, Valentine S, Hollander JE. Development and validation of a novel scar evaluation scale. Plast Reconstr Surg. 2007 Dec;120(7):1892-1897. doi: 10.1097/01.prs.0000287275.15511.10. PMID 18090752
- [Background] Quinn JV, Drzewiecki AE, Stiell IG, Elmslie TJ. Appearance scales to measure cosmetic outcomes of healed lacerations. Am J Emerg Med. 1995 Mar;13(2):229-31. doi: 10.1016/0735-6757(95)90100-0. PMID 7893315
- [Background] Gilbert L, Pogorzalek N, Jounda G, Barreau E. [Traumatic peri-ocular injuries: closing wounds using 2-octyl-cyanoacrylate medical glue]. J Fr Ophtalmol. 2009 May;32(5):341-7. doi: 10.1016/j.jfo.2009.03.024. Epub 2009 May 17. French. PMID 19769871
- [Background] Greene D, Koch RJ, Goode RL. Efficacy of octyl-2-cyanoacrylate tissue glue in blepharoplasty. A prospective controlled study of wound-healing characteristics. Arch Facial Plast Surg. 1999 Oct-Dec;1(4):292-6. doi: 10.1001/archfaci.1.4.292. PMID 10937118
- [Background] Handschel JG, Depprich RA, Dirksen D, Runte C, Zimmermann A, Kubler NR. A prospective comparison of octyl-2-cyanoacrylate and suture in standardized facial wounds. Int J Oral Maxillofac Surg. 2006 Apr;35(4):318-23. doi: 10.1016/j.ijom.2005.10.003. Epub 2005 Dec 20. PMID 16364595
- [Background] Shivamurthy DM, Singh S, Reddy S. Comparison of octyl-2-cyanoacrylate and conventional sutures in facial skin closure. Natl J Maxillofac Surg. 2010 Jan;1(1):15-9. doi: 10.4103/0975-5950.69151. PMID 22442543
- [Background] Hollander JE, Singer AJ, Valentine S, Henry MC. Wound registry: development and validation. Ann Emerg Med. 1995 May;25(5):675-85. doi: 10.1016/s0196-0644(95)70183-4. PMID 7741347